CLINICAL TRIAL: NCT04433091
Title: 2-Hydroxybenzylamine (2-HOBA) to Prevent Early Recurrence of Atrial Fibrillation After Catheter- Based Ablation
Brief Title: 2-Hydroxybenzylamine (2-HOBA) to Prevent Early Recurrence of Atrial Fibrillation After Catheter-based Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, M. Benjamin Shoemaker, Assoc Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 192520
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, randomized study. Eligible subjects will be randomized according to a permuted block scheme with a block size of balancing interval, varying randomly according to the outcome of a computer-generated random number. This ensures that the cumulative number of assignments to each treatment (2-HOBA or placebo) will be in balance after each block of assignments had been made. A statistician will design the randomization table and enable the randomization tool within REDCap. After a patient enrolls for the study, the study nurse will determine the treatment assignment using the randomization tool in REDCap.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant, care provider and investigator will all be blinded to the assigned treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2-HOBA (Active Comparator): 2-Hydroxybenzylamine(2-HOBA) 250 mg three tabs TID (po) for seven days prior to ablation and 28 days post ablation.
  Interventions: Drug: 2-Hydroxybenzylamine
- Placebo (Placebo Comparator): Placebo- three tabs TID (po) for seven days prior to ablation and 28 days post-ablation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2-Hydroxybenzylamine — 2-HOBA (2-Hydroxybenzlamine) 750mg will be given TID seven days prior to ablation and 28 days post ablation.
  Other Names: 2- HOBA
  Arms: 2-HOBA
Other: Placebo — Placebo will be given TID for seven days prior to ablation and 28 days post ablation.
  Arms: Placebo

SUMMARY:
The proposed studies will test this hypothesis by randomizing patients with AF to 2-HOBA or placebo 7 days prior to AF ablation to allow 2-HOBA to reach steady-state levels. We hypothesize that tissue injury from AF ablation causes a large release of ROS that react with lipids to generate IsoLGs (Figure 2). In the absence of 2-HOBA, IsoLGs will react within seconds to form IsoLG-macromolecule adducts in atrial tissue, promoting early recurrence of AF. In the presence of 2-HOBA, IsoLGs will rapidly react to form IsoLG-macromolecule adducts in atrial tissue, promoting early recurrence of AF. In the presence of 2-HOBA, IsoLG will preferentially bind to and therefore be inactivated by 2-HOBA thereby sparing injury to the atrial tissue caused by oxidative stress and its contribution to early recurrence of AF. Early recurrence of AF will be measured by ECGs that are recorded once per day by a smartwatch (Apple Watch, Apple Inc., Cupertino, CA) with additional ECGs recorded by the participant if they experience symptoms of AF, or if the smartwatch alerts the participant of a possible AF episode via its auto-detection AF monitoring algorithm. The Apple Watch's AF algorithm is based on sampling of heart rate and variability and will give an audible alarm if those parameters indicate a possible episode of AF. The smartwatch records a single-lead ECG if the participant touches the watch with their contralateral hand. The day and time of the episode is also stored by the smartwatch. At the end of the 28-day follow-up period, study personnel will review the stored ECGs. Blood will be drawn prior to ablation and on post-procedure Day 1 for measurement of IsoLG-adduct levels. DNA will be extracted to explore a pharmacogenomic interaction with haplotypes at the chromosome 4q25 AF risk locus, which: 1) is strongly associated with the development of AF and the early recurrence of AF after ablation27; and 2) has been reported to be a regulator of an anti-oxidant gene program in response to cardiac injury.

DETAILED DESCRIPTION:
The proposed double-blind, randomized, placebo-controlled trial of 2-HOBA in patients undergoing AF ablation is designed to address the following Specific Aims:

Specific Aim 1: To test the hypothesis that treatment with 2-HOBA reduces early recurrence of AF (clinical endpoint)

Specific Aim 2: To test the hypothesis that treatment with 2-HOBA reduces circulating levels of IsoLG-adducts (biochemical endpoint)

Specific Aim 3: To explore the idea that genetic variation at the 4q25 (PITX2) AF susceptibility locus modulates the clinical and biochemical response to 2-HOBA

ELIGIBILITY:
Inclusion Criteria:

* First time AF ablation with radiofrequency or cryo ablation
* Repeat AF ablation if the patient has persistent AF and ablation of non-pulmonary vein substrate is planned (e.g. posterior wall ablation, mitral or roof line, etc)
* Able to provide written, informed consent
* 22 years of age or older

Exclusion Criteria:

* Planned surgical or hybrid (surgical + catheter) ablation
* Amiodarone within past 3 months
* Use of oral steroids or colchicine
* Pro-inflammatory, rheumatologic disorder (e.g. RA, SLE, IBD, psoriasis, ankylosing spondylitis)
* NYHA Class III/IV Heart Failure
* LVEF <35%
* Active ischemia
* Hypertrophic Cardiomyopathy
* Cardiac or thoracic surgery within 6 months
* Expected life span < 1 year
* Creatinine clearance <30 ml/min
* Prior or planned heart transplantation
* Pregnant women
* Aspirin allergy
* Current use of MAO-I

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Shoemaker, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical, Nashville, Tennessee, United States

REFERENCES:
- [Derived] O'Neill MJ, Yoneda ZT, Crawford DM, Ye F, Ao M, Pitchford LM, Rathmacher JA, Murray KT, Akers WS, Roden DM, Michaud GF, Shoemaker MB. 2-Hydroxybenzylamine (2-HOBA) to prevent early recurrence of atrial fibrillation after catheter ablation: protocol for a randomized controlled trial including detection of AF using a wearable device. Trials. 2021 Aug 28;22(1):576. doi: 10.1186/s13063-021-05553-6. PMID 34454591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects will be identified through EPIC. The study team will approach the patient in person in Arrhythmia Clinic or by phone prior to AF ablation. Information describing the study, will be provided. The risks and benefits will be described along with potential treatment advances. Informed consent will be obtained with the option of phone consent with electronic signature.
Pre-assignment Details: 95 participants signed consent. 89 participants were randomized. 6 were withdrawn after enrollment and never randomized.
Period: Overall Study
Arm/Group | 2-HOBA | Placebo
Started | 46 | 43
Completed | 43 | 39
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawn . | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-HOBA | Placebo | Total
Number analyzed (Participants) | 43 | 39 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 51
  >=65 years | 16 | 15 | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 66] | 63 [57.5 to 70] | 63 [57 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 27 | 26 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 39 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 39 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 39 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Atrial Fibrillation
Description: Participants will wear a smartwatch linked to an iPhone to continually record heart rate, variability and detection of arrhythmias.
  Participants will record a daily ECG each morning upon waking via the watch. In addition, participants will be notified by the smartwatch of 1) detection of atrial fibrillation or atrial flutter, 2) persistent high HR (> 110 bpm) outside of exercise
Time Frame: Post-ablation through 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2-HOBA | Placebo
Number analyzed (Participants) | 43 | 39
Participants | 26 | 14

2. Secondary Outcome: The Change in IsoLG-adducts Levels From AF Pre-ablation to Post-procedure Day #1
Description: Circulating IsoLG adducts can be measured in the blood at different periods of time.
Time Frame: Pre-ablation and Post-procedure day #1
Population: This outcome required blood draw collections 1 day post ablation. During the Covid pandemic, this became impractical on approx. half the patients. IsoLG levels were only collected and analyzed on patients for whom blood samples were available.
Measure: Median (Inter-Quartile Range); unit: percentage of IsoLG in circ. monocytes
Arm/Group | 2-HOBA | Placebo
Number analyzed (Participants) | 23 | 22
percentage of IsoLG in circ. monocytes | 3.37 [.86 to 27.8] | 4.52 [.9 to 38.5]

3. Secondary Outcome: Exploratory Secondary Outcome
Description: AF burden obtained from smartwatch as defined by the percentage of time in AF compared to the time the smartwatch was worn.
Time Frame: 28 days post ablation
Population: The Apple Watch tracings were available to adjudicate recurrence in the final study cohort. However, burden required more data collection. Two of the participants were unable to provide the data. 1 participant refused.
  Outcome measure three part B required blood draw collections 1 day post ablation. During the Covid pandemic, this became impractical on ~half the patients. Outcome measure B (isoLG levels) were only collected and analyzed on patients for whom blood samples were available
Measure: Median (Inter-Quartile Range); unit: percentage of time in AF
Arm/Group | 2-HOBA | Placebo
Number analyzed (Participants) | 42 | 36
percentage of time in AF | 0 [0 to 0.007] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: First 28 days
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, only if it was considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion.
Arm/Group | 2-HOBA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/39
Other Adverse Events (participants affected / at risk) | 3/43 | 7/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2-HOBA (N=43) | Placebo (N=39)
nausea (Gastrointestinal disorders) | 3 | 5 — nausea
Headache (Nervous system disorders) | 0 | 2 — headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04433091/Prot_SAP_000.pdf